CLINICAL TRIAL: NCT06402825
Title: Follow-up of Children Born From a Randomized Controlled Trial Assessing a Preconception Lifestyle Intervention in Women With Obesity and Infertility
Brief Title: Obesity-fertility Cohort Study: Protocol for the Assessment of Children Aged 6-12 Years and Their Mothers
Status: Enrolling by invitation | Type: Observational
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Principal Investigator, Jean-Patrice Baillargeon, Associate Professor, Université de Sherbrooke
Other Study IDs: 2024-5150
Record Dates: First submitted 2024-04-23; First posted 2024-05-07 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-03

CONDITIONS: Obesity, Childhood; Lifestyle Intervention; Preconception Care
Keywords: Obesity; Maternal obesity; Healthy lifestyle; Preconception care; Fetal programming
MeSH Terms: conditions — Pediatric Obesity; Obesity; Pregnancy in Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Plasma, saliva
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Intervention: Children born from mothers who were allocated to the intervention group in the Obesity-Fertility study.
  Interventions: Behavioral: Fit-for-Fertility program
- Control: Children born from mothers who were allocated to the control group in the Obesity-Fertility study. Participants in the control group received standard care from the fertility clinic without delay.

INTERVENTIONS:
Behavioral: Fit-for-Fertility program — Women in the intervention group had to delay fertility treatments for 6 months and were offered the interdisciplinary lifestyle intervention, which was provided for a maximum of 18 months or until the end of a pregnancy that occurred. The lifestyle intervention consisted of individual meetings with a dietitian and a kinesiologist trained in motivational interviewing, combined with 12 educational group sessions during the first 6 months. Details of the lifestyle intervention are presented in the previously published protocol (Duval et al., 2015).
  Groups: Intervention

SUMMARY:
Maternal preconception obesity and adverse gestational metabolic health increase the risk of childhood obesity in offspring. A group of investigators from Université de Sherbrooke therefore developed a lifestyle intervention starting during preconception in women with obesity and infertility, which was evaluated with the Obesity-Fertility randomized controlled trial (RCT). The present study will assess children who were born in the Obesity-Fertility RCT and are now aged 6-10 years old. The objective of this study is to evaluate the effect of a lifestyle intervention during preconception and pregnancy on adiposity and cardiometabolic parameters in offspring compared to those born to mothers who did not have access to the lifestyle intervention. The hypothesis being that, at the age of 6-10 years old, children born to mothers who were in the intervention group have more favorable measurements of body composition and certain metabolic and/or inflammatory blood markers than those born to control mothers.

Participants in the Obesity-Fertility RCT were women with obesity and infertility recruited at the Centre hospitalier universitaire de Sherbrooke (CHUS) fertility clinic. They were randomly allocated to the control group, which followed standard care, or to the intervention group, which received a lifestyle intervention alone for 6 months, and then in combination with fertility treatments. Those who have given birth to a single child will be invited to participate in this follow-up study with their child. During the research visit, medical history, anthropometry, body composition, lifestyle, physical fitness level, and blood or saliva markers of cardiometabolic health will be assessed for both mothers and children.

This study will provide new evidence on the impact of targeting lifestyle habits during preconception on the health of children and their mothers 6-10 years later; and the potential of such interventions to counteract the intergenerational transmission of obesity.

DETAILED DESCRIPTION:
INTRODUCTION: Maternal preconception obesity and adverse gestational metabolic health increase the risk of childhood obesity in offspring. A group of investigators from Université de Sherbrooke therefore developed a lifestyle intervention starting during preconception in women with obesity and infertility, which was evaluated with the Obesity-Fertility randomized controlled trial (RCT) registered at ClinicalTrials.gov (NCT01483612). The present study will assess children who were born in the Obesity-Fertility RCT and are now aged 6-10 years old. The objective of this study is to evaluate the effect of a lifestyle intervention during preconception and pregnancy on adiposity and cardiometabolic parameters in offspring compared to those born to mothers who did not have access to the lifestyle intervention.

METHODS AND ANALYSIS: Participants in the Obesity-Fertility RCT were women with obesity and infertility recruited at the CHUS fertility clinic between January 2012 and August 2018. They were randomly allocated to the control group, which followed standard care, or to the intervention group, which received a lifestyle intervention alone for 6 months, and then in combination with fertility treatments. Those who have given birth to a single child will be invited to participate in this follow-up study with their child. This study will take place from October 2023 to September 2024, when the child will be 6-10 years old. During the research visit, medical history, anthropometry, body composition, lifestyle, physical fitness level, and blood or saliva markers of cardiometabolic health will be assessed for both mothers and children. Of the 130 women who participated in the Obesity-Fertility RCT, 53 mother-child dyads are potentially eligible for this follow-up study. Comparisons between groups will be performed using appropriate unpaired tests and adjusted for potential confounders using multiple regression models.

ETHICS AND DISSEMINATION: The study has been approved by the Institutional Research Ethics Review Boards of the CHUS. The results will be widely disseminated to the scientific community as well as to relevant health professionals and the general public.

IMPACT: This study will provide new evidence on the impact of targeting lifestyle habits during preconception on the health of children and their mothers 6-10 years later; and the potential of such interventions to counteract the intergenerational transmission of obesity.

ELIGIBILITY:
Inclusion Criteria:

* Offsprings of women who were randomized in the Obesity-Fertility study known to have been conceived within 18 months following randomization of their mothers from a singleton pregnancy.

Exclusion Criteria:

* Children having a disease or taking a medication that has a major impact on weight, anthropometry, lifestyle habits or functional capacity (e.g., congenital heart disease, functional disability, severe asthma, regular use of glucocorticoids, etc.).

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children born from mothers who participated in the Obesity-Fertility study. Those mother were recruited between 2012 and 2018 at the fertility clinic of the Centre hospitalier universitaire de Sherbrooke. To be included in the study, they had to be aged between 18 and 40 years and living with infertility and obesity, or overweight if they had polycystic ovary syndrome (PCOS). Women were excluded if they had undergone or were planning bariatric surgery, or if natural conception was impossible or unlikely (such as both fallopian tubes blocked or severe male factor).
Sampling Method: Non-Probability Sample
Enrollment: 47 (Estimated)
Dates: Start 2023-11-13 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Anthropometrics - BMI z score (child) | Once, between October 2023 and September 2024 (11 months), which is 6 to 10 years after the child's birth.
  BMI Z-score adjusted for age and sex calculated according to World Health Organization reference values (AnthroPlus software, version 1.0, last updated September 17, 2014)

SECONDARY OUTCOMES:
Anthropometrics - Waist circumference | Once, between October 2023 and September 2024 (11 months), which is 6 to 10 years after the child's birth.
  Measured at the highest point of the iliac crests according to the National Institutes of Health (NIH) method to the nearest 0.1 cm with a flexible tape
Anthropometrics - Waist-to-height ratio (child) | Once, between October 2023 and September 2024 (11 months), which is 6 to 10 years after the child's birth.
  Calculated from the child's waist circumference (cm) and height (cm).
Body composition measured by dual-energy X-ray absorptiometry | Once, between October 2023 and September 2024 (11 months), which is 6 to 10 years after the child's birth.
  Fat and lean body mass, ratio
Lifestyle - Self-reported physical activity by GSLTPAQ (child) | Once, between October 2023 and September 2024 (11 months), which is 6 to 10 years after the child's birth.
  Godin-Shephard Leisure-Time Physical Activity Questionnaire (GSLTPAQ) measures frequency and intensity of physical activity practiced by the child during the past seven days
Lifestyle - Self-reported physical activity level (mother) | Once, between October 2023 and September 2024 (11 months), which is 6 to 10 years after the child's birth.
  Questionnaire adapted from the 2009 Canadian Community Health Survey of Statistics Canada
Lifestyle - Number of steps per day measured by Fitbit (child) | Once, over a one-week period, between October 2023 and September 2024 (11 months), which is 6 to 10 years after the child's birth.
  Fitbit wristband monitor worn for seven consecutive days
Lifestyle - Minutes per day of physical activity measured by Fitbit (child) | Once, over a one-week period, between October 2023 and September 2024 (11 months), which is 6 to 10 years after the child's birth.
  Fitbit wristband monitor worn for seven consecutive days
Lifestyle - Dietary behaviours by CTFEQr17 (child) | Once, between October 2023 and September 2024 (11 months), which is 6 to 10 years after the child's birth.
  French version of the Child Three-Factor Eating Questionnaire (CTFEQr17)
Lifestyle - Food intake (child) | Three dietary recall, over a period of four weeks, between October 2023 and September 2024 (11 months), which is 6 to 10 years after the child's birth.
  Online 24-hour dietary recall survey developed by Laval University
Lifestyle - Eating habits (mother) | Once, between October 2023 and September 2024 (11 months), which is 6 to 10 years after the child's birth.
  Questionnaire adapted from the 2009 Canadian Community Health Survey of Statistics Canada
Physical fitness level - Cardiorespiratory fitness (child) | Once, between October 2023 and September 2024 (11 months), which is 6 to 10 years after the child's birth.
  Maximal exertion test using the McMaster protocol
Physical fitness level - Grip strength (child) | Once, between October 2023 and September 2024 (11 months), which is 6 to 10 years after the child's birth.
  Hand dynamometer (kg)
Physical fitness level - Functional capacity (mother) | Once, between October 2023 and September 2024 (11 months), which is 6 to 10 years after the child's birth.
  Six-minute walk test
Cardiometabolic health - Systolic and diastolic blood pressure | Once, between October 2023 and September 2024 (11 months), which is 6 to 10 years after the child's birth.
  Arm cuff appropriate for the arm size (mmHg)
Cardiometabolic health - Systolic and diastolic blood pressure Z-scores (child) | Once, between October 2023 and September 2024 (11 months), which is 6 to 10 years after the child's birth.
  Age-, sex- and height-adjusted Z-scores from normative tables from the American Academy of Pediatrics Pediatric Reference Guidelines
Cardiometabolic health - Heart rate | Once, between October 2023 and September 2024 (11 months), which is 6 to 10 years after the child's birth.
  Arm cuff appropriate for the arm size (bpm)
Cardiometabolic health - Total cholesterol (TC) | Once, between October 2023 and September 2024 (11 months), which is 6 to 10 years after the child's birth.
  Fasting levels
Cardiometabolic health - Triglycerides | Once, between October 2023 and September 2024 (11 months), which is 6 to 10 years after the child's birth.
  Fasting levels
Cardiometabolic health - High-density lipoprotein (HDL) cholesterol | Once, between October 2023 and September 2024 (11 months), which is 6 to 10 years after the child's birth.
  Fasting levels
Cardiometabolic health - Low-density lipoprotein (LDL) cholesterol | Once, between October 2023 and September 2024 (11 months), which is 6 to 10 years after the child's birth.
  Fasting levels
Cardiometabolic health - Cholesterol ratio | Once, between October 2023 and September 2024 (11 months), which is 6 to 10 years after the child's birth.
  Fasting levels of TC divide by fasting levels of HDL

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Patrice Baillargeon, MD, Principal Investigator — Université de Sherbrooke
Locations (1):
- Centre hospitalier universitaire de Sherbrooke, Sherbrooke, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Duval K, Langlois MF, Carranza-Mamane B, Pesant MH, Hivert MF, Poder TG, Lavoie HB, Ainmelk Y, St-Cyr Tribble D, Laredo S, Greenblatt E, Sagle M, Waddell G, Belisle S, Riverin D, Jean-Denis F, Belan M, Baillargeon JP. The Obesity-Fertility Protocol: a randomized controlled trial assessing clinical outcomes and costs of a transferable interdisciplinary lifestyle intervention, before and during pregnancy, in obese infertile women. BMC Obes. 2015 Dec 1;2:47. doi: 10.1186/s40608-015-0077-x. eCollection 2015. PMID 26635965
- [Derived] Thibodeau A, Jean-Denis F, Harnois-Leblanc S, Perron P, Mathieu ME, Dallaire F, Morisset AS, Brochu M, Baillargeon JP. Obesity-fertility cohort study: protocol for the assessment of children aged 6-12 years and their mothers. BMJ Open. 2025 Apr 17;15(4):e091140. doi: 10.1136/bmjopen-2024-091140. PMID 40246570